CLINICAL TRIAL: NCT03028649
Title: The Effect of β-hydroxy-β-methylbutyrate (HMB) Supplementation on Physical Capacity and Body Composition in Trained Athletes
Brief Title: The Effect of β-hydroxy-β-methylbutyrate Supplementation on Physical Capacity and Body Composition in Trained Athletes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Collaborators: Poznan University of Life Sciences (Other); National Science Centre, Poland (Other Government)
Responsible Party: Principal Investigator, Krzysztof Durkalec-Michalski, Assistant Professor, Poznan University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NN312262340
Record Dates: First submitted 2017-01-11; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Sport; Supplements; Supplementation
Keywords: β-hydroxy-β-methylbutyric acid; Sport supplements; Training support; Adaptation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- β-hydroxy-β-methylbutyrate (HMB) (Experimental): Group taking oral supplementation with calcium salt of β-hydroxy-β-methylbutyric acid produced by Olimp Laboratories. A single capsule contained 1250 mg Ca-HMB, which corresponds to 1000 mg of β-hydroxy-β-methylbutyrate.
  Interventions:
  The experimental procedure for each athlete included a 12-week HMB supplementation - 3 capsules of the assigned preparation a day in 3 doses: upon waking, immediately after training, and before sleep. On non-training days, the participants were instructed to consume one serving with each of three separate meals throughout the day.
  Between the 12-week HMB and PLA or a PLA and HMB treatment, a 10-day washout period was introduced.
  Interventions: Dietary Supplement: β-hydroxy-β-methylbutyrate and a placebo supplementation
- Placebo (maltodextrin) (Placebo Comparator): Group taking oral supplementation with placebo (maltodextrin). A single capsule contained 1000 mg of maltodextrin.
  Interventions:
  The experimental procedure for each athlete included a 12-week placebo administration - 3 capsules of the assigned preparation a day in 3 doses: upon waking, immediately after training, and before sleep. On non-training days, the participants were instructed to consume one serving with each of three separate meals throughout the day.
  Between the 12-week HMB and PLA or a PLA and HMB treatment, a 10-day washout period was introduced.
  Interventions: Dietary Supplement: β-hydroxy-β-methylbutyrate and a placebo supplementation

INTERVENTIONS:
Dietary Supplement: β-hydroxy-β-methylbutyrate and a placebo supplementation

SUMMARY:
The purpose of this study was to verify the effect of 12-week with β-hydroxy-β-methylbutyrate (HMB) and a placebo (PLA) supplementation on body composition, anaerobic and aerobic capacity, as well as concentrations of the selected biochemical blood markers in trained athletes, in a randomised, double-blind, placebo-controlled crossover trial.

DETAILED DESCRIPTION:
The effect of HMB supplementation is of great interest in sport. In view of the inconclusive character of the results of the studies conducted to date and of a relatively low number of studies investigating the effectiveness of HMB supplementation over a longer period on a large population of trained athletes, the aim of this study was to verify the effect of 12-week with HMB and a placebo supplementation on body composition, anaerobic and aerobic capacity, as well as concentrations of the selected biochemical blood markers in trained athletes, in a randomised, double-blind, placebo-controlled crossover trial.

ELIGIBILITY:
Inclusion Criteria:

* written consent to participate,
* male
* a current medical clearance to practice sports,
* training experience: at least 5 years,
* minimum of 6 workout sessions a week (minimum 3 in the practiced sports discipline).

Exclusion Criteria:

* current injury,
* any health-related contraindication,
* declared general feeling of being unwell,
* unwilling to follow the study protocol.

Ages: 17 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2010-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Changes of body composition indices after HMB supplementation | Baseline and after 12 weeks
  Analysis of the fat mass and fat free mass
Changes of body composition indices after placebo treatment | Baseline and after 12 weeks
  Analysis of the fat mass and fat free mass
Changes of aerobic capacity after HMB supplementation | Baseline and after 12 weeks
Changes of aerobic capacity after placebo treatment | Baseline and after 12 weeks
Changes of anaerobic capacity after HMB supplementation | Baseline and after 12 weeks
Changes of anaerobic capacity after placebo treatment | Baseline and after 12 weeks
Changes of creatine kinase and lactate dehydrogenase activity in blood after HMB supplementation | Baseline and after 12 weeks
Changes of creatine kinase and lactate dehydrogenase activity in blood after placebo treatment | Baseline and after 12 weeks
Changes of testosterone, cortisol and lactate levels in blood after HMB supplementation | Baseline and after 12 weeks
Changes of testosterone, cortisol and lactate levels in blood after placebo treatment | Baseline and after 12 weeks

SECONDARY OUTCOMES:
Statistical evaluation of the significance of differences between the changes in body composition (fat mass and fat free mass) | 1 year
Statistical evaluation of the significance of differences between the changes in aerobic capacity indices | 1 year
Statistical evaluation of the significance of differences between the changes in anaerobic capacity indices | 1 year
Statistical evaluation of the significance of differences between the changes in creatine kinase and lactate dehydrogenase activity and testosterone, cortisol and lactate levels in blood | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jan Jeszka, Professor, Study Chair — Department of Hygiene and Human Nutrition, Poznan University of Life Sciences, Poznan, Poland
Locations (1):
- Poznan University of Life Sciences, ul.Wojska Polskiego 31, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Shared data will be exclusively related to the level recorded indicators (body composition, aerobic and anaerobic capacity indicators, levels of biochemical markers), without personal data. The data obtained will be attached to scientific publications, depending on the requirements of the journal